CLINICAL TRIAL: NCT00325247
Title: Efficacy of Short Course Zinc Therapy (5 vs 10 d) With 20 mg Elemental Zinc Daily in the Treatment of Acute Diarrhoea: A Double-blind Individually Randomized Controlled Community Trial.
Brief Title: Efficacy of Zinc Therapy in Acute Diarrhoea in Young Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2004-018
Record Dates: First submitted 2006-05-11; First posted 2006-05-12 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2006-05

CONDITIONS: Acute Watery Diarrhoea
Keywords: ZINC SUPPLEMENTATION; ACUTE DIARRHOEA; UNDER FIVE CHILDREN; RURAL BANGLADESH
MeSH Terms: interventions — Zinc

INTERVENTIONS:
Drug: ZINC

SUMMARY:
Diarrhoea continues to be a major cause of mortality and morbidity in young children especially in many developing countries. Although the mortality burden of diarrhoea has substantially reduced, the morbidity pattern remained almost unchanged. Recent randomized controlled supplementation trials in developing countries have consistently shown that zinc has the potential to reduce the duration of diarrhoea as well as has preventive effect on childhood diarhroea in subsequent months. Currently, international health agencies recommend zinc as an important adjunct therapy to treat diarrhoea in developing countries where zinc deficiency is highly prevalent and diet is poor in zinc.

The recommendation is to provide 20 mg elemental zinc daily for 10 days during each episode of diarrhoea.

This study aims at evaluating the relative efficacy of two length of 20 mg zinc therapy (5 vs 10 days) during acute diarrhoea in a rural community in a community-based individually randomized placebo-controlled trial with 20 mg zinc daily and will be conducted in seven villages in the ICDDR,B Matlab study area.

The study will require 2050 acute dirrhoeal episodes to be treated who will be randomly allocated to one of the two treatment schedules (20 mg of zinc daily for 5 or 10 days). Children who will be allocated to the shorter duration therapy will receive placebo for the remaining days to complete 10-day treatment. Female Field Workers (FFWs) will conduct diarrhoea surveillance and administer zinc daily at home. Data will be analyzed using appropriate statistical procedure.

Findings of this study will be immensely valuable for deciding recommendation for the duration of zinc therapy in the management of acute diarrhoea in young children and will have profound programmatic and policy implications for scaling up zinc intervention in the community.

DETAILED DESCRIPTION:
The proposed study will use a prospective, double-blind, randomized design in which all study children with diarrhoea will receive zinc treatment for the first 5 days and then they will receive either zinc or a placebo for the second 5 days of the 10 day course according to random allocation to evaluate the efficacy of shorter course of zinc treatment (5 days vs 10 days) during diarrhoea in children less than 5 years of age. Children with diarrhoea will be detected through routine daily surveillance by trained Female Field Worker (FFW) in the study area and will be enrolled into the study soon after detection and the informed consent of the parent is obtained. Zinc will be administered daily by FFWs as 20 mg elemental zinc as single dose for 5 or 10 days. Dispersible zinc tablets in blister pack produced by Nutriset® used in the national zinc scaling up project will be used for the study. The placebo will also be dispersible tablets identical and undistinguishable from zinc tablet in terms of appearance, colour, taste and flavour will be obtained from the same manufacturer. The first episode of a child will be treated as part of this study although children will be encouraged to take zinc if s/he develops diarrhoea during the study period. The dose is about double the Recommended Daily Allowance (RDA) for the children which has been chosen considering the poor zinc status of the children to be included and replenishment of possible loss of zinc during diarrhoeal episode and also to be consistent with the current recommendation in the zinc scaling up initiative. Outcome will be assessed daily during routine visit using a precoded questionnaire. Although all the children will receive zinc treatment for one of the two durations, ones who will be randomly assigned to shorter duration (5 day) will receive zinc for the first 5 days and then placebo for the rest of the days to complete 10 days intake.

ELIGIBILITY:
Inclusion Criteria:

1. Children less than 5 years with acute watery diarrhoea less than 48 h of duration
2. No medication received other than ORS or home solution
3. Absence of complication or co-morbidities.
4. Absence of severe dehydration

Exclusion Criteria:

1. Age greater than 5 years
2. Diarrhoea more than 48 h duration
3. Unable to eat or drink
4. Already received multiple treatment including zinc
5. Presence of co-morbidities
6. Severe dehydration

Ages: 1 Month to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2050 (Estimated)
Dates: Start 2005-02; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Preventive effect of zinc therapy on diarrhoea during the subsequent three month 14 days of enrollment
Assess the acceptability of zinc therapy during diarrhoea in young children.

SECONDARY OUTCOMES:
Compare the duration of current episode in two groups receiving 5 d vs 10 d zinc.
Compare the proportion of children developing prolonged (>10 d) or persistent diarrheoa (>14 d).

CONTACTS AND LOCATIONS:
Overall Officials: Dewan S Alam, PhD, Principal Investigator — ICDDR,B: Centre for Health and Population Research
Locations (1):
- ICDDR,B, Dhaka, Bangladesh

REFERENCES:
- [Derived] Alam DS, Yunus M, El Arifeen S, Chowdury HR, Larson CP, Sack DA, Baqui AH, Black RE. Zinc treatment for 5 or 10 days is equally efficacious in preventing diarrhea in the subsequent 3 months among Bangladeshi children. J Nutr. 2011 Feb;141(2):312-5. doi: 10.3945/jn.110.120857. Epub 2010 Dec 8. PMID 21147907